CLINICAL TRIAL: NCT02046317
Title: Trial of Ultrasound Guided Femoral Nerve Block on Isolated Femur Fracture Using Echo Friendly Needles
Acronym: TUFFEN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No further enrolled patients, Primary researcher left the institution
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Carlos Roldan, Associate Professor - Emergency Medicine, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-11-0035
Record Dates: First submitted 2013-12-17; First posted 2014-01-27 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Echogenic needle (Experimental): The experimental arm will receive ultrasound-guided femoral nerve block using echogenic needles, which are micro laser etched near the tip to reflect sound waves back to the transducer and make the tip visible.
  Interventions: Drug: Femoral Nerve Block; Device: Echogenic needle; Device: Ultrasound
- Standard of care needle (Active Comparator): The control group will receive ultrasound-guided femoral nerve block using standard of care needles.
  Interventions: Drug: Femoral Nerve Block; Device: Standard of care needle; Device: Ultrasound

INTERVENTIONS:
Drug: Femoral Nerve Block — Femoral Nerve Block for isolated femur fractures
Device: Echogenic needle — The experimental arm will receive ultrasound-guided femoral nerve block using echogenic needles, which are micro laser etched near the tip to reflect sound waves back to the transducer and make the tip visible.
  Arms: Echogenic needle
Device: Standard of care needle — The control group will receive ultrasound-guided femoral nerve block using standard of care needles.
  Arms: Standard of care needle
Device: Ultrasound — The experimental arm will receive ultrasound-guided femoral nerve block using echogenic needles, which are micro laser etched near the tip to reflect sound waves back to the transducer and make the tip visible.
  The control group will receive ultrasound-guided femoral nerve block using standard of care needles.

SUMMARY:
This study aims to determine if there is any difference in the success rate of ultra-sound guided femoral nerve block performed with an echogenic needle versus a standard needle.

DETAILED DESCRIPTION:
To date, the published information regarding ultrasound guided femoral nerve blocks (FNB) using echo friendly needle is very limited. More so, there is even less information regarding ultrasound guided nerve blocks using echogenic versus standard of care needles.

This study hopes to add to the general knowledge of pain management in the emergency department (ED) setting and provide a unique perspective on ultrasound-guided techniques using echogenic needles to enhance accuracy and success rate of nerve blocks in ED patients.

The study design will have two comparative arms; in both arms we use the same local anesthetic which is Bupivacaine 0.25% with epinephrine; in all cases a total of 15 mL will be injected around the femoral nerve. Once identified with ultrasound, 5 ml will be injected at lateral, medial, and posterior aspect of the nerve. The experimental arm will receive an FNB using an echogenic needle; and the control group will receive an FNB using standard of care needles.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the emergency department (ED) with isolated femur fracture (no other injuries)
* Patients who are cognitively alert and are able to verbalize their pain using a visual analog scale (VAS)
* Patients who are mentally competent to consent for the study
* Patients who can communicate in English or Spanish

Exclusion Criteria:

* Gestation
* Prisoners
* Patients who cannot communicate in English or in Spanish
* Patients who have other significant injuries besides a femur fracture
* Patients who are cognitively impaired and/or unable to verbalize their pain using a visual analog scale (VAS)
* Patients with allergies to local anesthetics
* Patients with severe liver disease
* Patients with existing peripheral neuropathies in the affected limb
* Patients with history of complications from previous femoral blocks
* Patients with contraindications for needle insertion at inguinal area
* Local signs of infection
* Patient on anticoagulants and/or with history of coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos J Roldan, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Memorial Hermann Hospital Texas Medical Center, Houston, Texas

REFERENCES:
- [Background] Beaudoin FL, Nagdev A, Merchant RC, Becker BM. Ultrasound-guided femoral nerve blocks in elderly patients with hip fractures. Am J Emerg Med. 2010 Jan;28(1):76-81. doi: 10.1016/j.ajem.2008.09.015. PMID 20006206
- [Background] Bijur P, Berard A, Nestor J, Calderon Y, Davitt M, Gallagher EJ. No racial or ethnic disparity in treatment of long-bone fractures. Am J Emerg Med. 2008 Mar;26(3):270-4. doi: 10.1016/j.ajem.2007.05.010. PMID 18358935
- [Background] Brull R, Perlas A, Chan VW. Ultrasound-guided peripheral nerve blockade. Curr Pain Headache Rep. 2007 Feb;11(1):25-32. doi: 10.1007/s11916-007-0018-6. PMID 17214918
- [Background] Deam RK, Kluger R, Barrington MJ, McCutcheon CA. Investigation of a new echogenic needle for use with ultrasound peripheral nerve blocks. Anaesth Intensive Care. 2007 Aug;35(4):582-6. doi: 10.1177/0310057X0703500419. PMID 18020079
- [Background] Fletcher AK, Rigby AS, Heyes FL. Three-in-one femoral nerve block as analgesia for fractured neck of femur in the emergency department: a randomized, controlled trial. Ann Emerg Med. 2003 Feb;41(2):227-33. doi: 10.1067/mem.2003.51. PMID 12548273
- [Background] Haddad FS, Williams RL. Femoral nerve block in extracapsular femoral neck fractures. J Bone Joint Surg Br. 1995 Nov;77(6):922-3. PMID 7593107
- [Background] Iamaroon A, Raksakietisak M, Halilamien P, Hongsawad J, Boonsararuxsapong K. Femoral nerve block versus fentanyl: Analgesia for positioning patients with fractured femur. Local Reg Anesth. 2010;3:21-6. doi: 10.2147/lra.s8600. Epub 2010 Mar 25. PMID 22915864
- [Background] Lee JS, Hobden E, Stiell IG, Wells GA. Clinically important change in the visual analog scale after adequate pain control. Acad Emerg Med. 2003 Oct;10(10):1128-30. doi: 10.1111/j.1553-2712.2003.tb00586.x. PMID 14525749
- [Background] Marhofer P, Chan VW. Ultrasound-guided regional anesthesia: current concepts and future trends. Anesth Analg. 2007 May;104(5):1265-9, tables of contents. doi: 10.1213/01.ane.0000260614.32794.7b. PMID 17456684
- [Background] Marhofer P, Schrogendorfer K, Wallner T, Koinig H, Mayer N, Kapral S. Ultrasonographic guidance reduces the amount of local anesthetic for 3-in-1 blocks. Reg Anesth Pain Med. 1998 Nov-Dec;23(6):584-8. doi: 10.1016/s1098-7339(98)90086-4. PMID 9840855
- [Background] Marhofer P, Schrogendorfer K, Koinig H, Kapral S, Weinstabl C, Mayer N. Ultrasonographic guidance improves sensory block and onset time of three-in-one blocks. Anesth Analg. 1997 Oct;85(4):854-7. doi: 10.1097/00000539-199710000-00026. PMID 9322469
- [Background] Moher D, Dulberg CS, Wells GA. Statistical power, sample size, and their reporting in randomized controlled trials. JAMA. 1994 Jul 13;272(2):122-4. PMID 8015121
- [Background] Mutty CE, Jensen EJ, Manka MA Jr, Anders MJ, Bone LB. Femoral nerve block for diaphyseal and distal femoral fractures in the emergency department. Surgical technique. J Bone Joint Surg Am. 2008 Oct;90 Suppl 2 Pt 2:218-26. doi: 10.2106/JBJS.H.00314. PMID 18829935
- [Background] Saygi B, Ozkan K, Eceviz E, Tetik C, Sen C. Skin traction and placebo effect in the preoperative pain control of patients with collum and intertrochanteric femur fractures. Bull NYU Hosp Jt Dis. 2010;68(1):15-7. PMID 20345356
- [Background] Terrell KM, Hui SL, Castelluccio P, Kroenke K, McGrath RB, Miller DK. Analgesic prescribing for patients who are discharged from an emergency department. Pain Med. 2010 Jul;11(7):1072-7. doi: 10.1111/j.1526-4637.2010.00884.x. PMID 20642733
- [Background] Tondare AS, Nadkarni AV. Femoral nerve block for fractured shaft of femur. Can Anaesth Soc J. 1982 May;29(3):270-1. doi: 10.1007/BF03007129. PMID 7074406

RESULTS

PARTICIPANT FLOW:
Groups:
- Echogenic Needle: The experimental arm will receive ultrasound-guided femoral nerve block using echogenic needles, which are micro laser etched near the tip to reflect sound waves back to the transducer and make the tip visible.
  Femoral Nerve Block: Femoral Nerve Block for isolated femur fractures
  Echogenic needle: The experimental arm will receive ultrasound-guided femoral nerve block using echogenic needles, which are micro laser etched near the tip to reflect sound waves back to the transducer and make the tip visible.
  Ultrasound: The experimental arm will receive ultrasound-guided femoral nerve block using echogenic needles, which are micro laser etched near the tip to reflect sound waves back to the transducer and make the tip visible.
  The control group will receive ultrasound-guided femoral nerve block using standard of care needles.
- Standard of Care Needle: The control group will receive ultrasound-guided femoral nerve block using standard of care needles.
  Femoral Nerve Block: Femoral Nerve Block for isolated femur fractures
  Standard of care needle: The control group will receive ultrasound-guided femoral nerve block using standard of care needles.
  Ultrasound: The experimental arm will receive ultrasound-guided femoral nerve block using echogenic needles, which are micro laser etched near the tip to reflect sound waves back to the transducer and make the tip visible.
  The control group will receive ultrasound-guided femoral nerve block using standard of care needles.
Period: Overall Study
Arm/Group | Echogenic Needle | Standard of Care Needle
Started | 4 | 8
Completed | 4 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Echogenic Needle | Standard of Care Needle | Total
Number analyzed (Participants) | 4 | 8 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.25 (35.55) | 66.88 (13.70) | 61.67 (22.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Patient Pain Level
Description: Pain level will be measured on a numeric visual analogue scale of 0-10 with 0 being no pain and 10 being the worst pain ever.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Echogenic Needle | Standard of Care Needle
Number analyzed (Participants) | 4 | 8
units on a scale | 7.50 (2.38) | 8.00 (2.07)

2. Primary Outcome: Patient Pain Level
Description: as for outcome 1
Time Frame: 60 minutes after initial femoral block
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Echogenic Needle | Standard of Care Needle
Number analyzed (Participants) | 4 | 8
units on a scale | 1.25 (2.50) | 3.75 (2.92)

ADVERSE EVENTS:
Time Frame: Length of stay in Emergency Department (about 5 hours)
Arm/Group | Echogenic Needle | Standard of Care Needle
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 0/4 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes